CLINICAL TRIAL: NCT01809431
Title: Optimizing Outcomes in Women With Gestational Diabetes Mellitus and Their Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0486; 1R21DK092750-01A1 (NIH)
Record Dates: First submitted 2013-03-10; First posted 2013-03-12 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2015-06

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; women; infants; blood glucose; weight; adiposity; health behaviors; self-efficacy
MeSH Terms: conditions — Diabetes, Gestational; Body Weight; Obesity; Health Behavior | interventions — Methods; Nutrition Assessment; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): Breastfeeding, progression to type 2 diabetes, nutrition, and exercise education, coping skills training, exercise training, a home-based exercise program and educational and motivational text messaging.
  Interventions: Behavioral: Intervention
- Wait-listed control group (No Intervention): Wait-listed control group receive usual care delivered by their health care provider and after completion of their time in the study they are offered the intervention

INTERVENTIONS:
Behavioral: Intervention — Using a two-group, repeated measures experimental design, this proposed study will test a 14-week intensive intervention on the benefits of breastfeeding, understanding gestational diabetes and risk of progression to prediabetes and type 2 diabetes, nutrition and exercise education, coping skills training, and physical activity (Phase I) and 3 months of continued monthly contact (Phase II) to help overweight women diagnosed with gestational diabetes improve metabolic, clinical, weight, adiposity, health behaviors and self-efficacy.
  Other Names: breastfeeding education; progression to prediabetes and type 2 diabetes education; nutrition education; exercise education; coping skills training; exercise training; home-based exercise program; educational and motivational text messaging
  Arms: intervention

SUMMARY:
The purpose of this study is to determine whether a 14 week intervention is successful in improving outcomes for women with gestational diabetes mellitus and their infants.

DETAILED DESCRIPTION:
Women who are diagnosed with gestational diabetes are at increased risk for developing prediabetes and type 2 diabetes. To date, there have been few interdisciplinary interventions that target predominantly ethnic minority low-income women diagnosed with gestational diabetes. Programs are needed that intervene in the prenatal period to teach women the importance of breastfeeding to improve metabolic control and infant health and continue after birth to promote improved nutrition and exercise patterns and weight loss. Using a two-group, repeated measures experimental design, this proposed study will test a 14-week intensive intervention on the benefits of breastfeeding, understanding gestational diabetes and risk of progression to prediabetes and type 2 diabetes, nutrition and exercise education, coping skills training, and physical activity (Phase I) and 3 months of continued monthly contact (Phase II) to help overweight women diagnosed with gestational diabetes improve metabolic, clinical, weight, adiposity, health behaviors and self-efficacy. Trends in breastfeeding duration and intensity, maternal infant feeding behavior, infant growth trajectory (weight-for-length) will also be measured. A total of 100 African American, bilingual Hispanic, and non-Hispanic White women diagnosed with gestational diabetes will be inducted and randomized by site to either the experimental or wait-list control group. Data will be collected at Time 1 (Baseline at 22-36 weeks pregnant), Time 2 (6 weeks postpartum), Time 3 (4 months postpartum and completion of Phase I), Time 4 (7 months postpartum and completion of Phase II), and Time 5 (10 months postpartum and after 3 months on their own). Primary maternal outcomes will include fasting blood glucose and weight (BMI). Secondary maternal outcomes will include clinical outcomes (oral glucose tolerance test, insulin levels, Homeostasis Model Assessment calculation, Hemoglobin A1c, complete lipid panel, and blood pressure); adiposity (waist circumference, triceps and subscapular skin folds); health behaviors (Health Promoting Lifestyle Profile II, Adult Health Behavior Survey, and Accelerometry for 7 days); and self-efficacy (Eating Self-Efficacy, Exercise Self-Efficacy Scale, and Breastfeeding Self-Efficacy Scale). Infant outcomes will include data on weight status (weight-for-length) and breastfeeding (weeks until stopped breastfeeding, weeks exclusively breastfed, and intensity of breastfeeding). Data analysis will include analysis of field notes, post-intervention interviews, and recruitment and retention efforts. Linear mixed-effects random coefficients models will be constructed to measure the effects of the intervention compared to the wait-list control group. Increasing breastfeeding and decreasing overweight in postpartum women who were diagnosed with gestational diabetes may both improve maternal glucose homeostasis and weight and stabilize infant growth trajectory, reducing the burden of metabolic disease across two generations.

ELIGIBILITY:
Inclusion Criteria:

* Women between 22-36 weeks of pregnancy who are diagnosed with GDM
* A diagnosis of GDM during the current pregnancy by two or more 100g Oral Glucose Tolerance Test (OGTT) values exceeding established thresholds (fasting 95, 1h 180, 2h 155, 3h 140 mg/dL)
* Age 18-45 years old
* A pre-pregnancy body mass index > 25kg/m2

  * Ability to read and write in English
  * Willingness to consent for themselves and their infant

Exclusion Criteria:

* They have a A1c ≥ 6.5 mg/dL (Type 2 diabetes)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
fasting blood glucose | Baseline to 10 months postpartum
  Change in fasting blood glucose in mothers
weight (body mass index) | Baseline to 10 months postpartum
  Change in weight (body mass index)in mothers

SECONDARY OUTCOMES:
oral glucose tolerance test | Baseline to 10 months postpartum
  Change in oral glucose tolerance test in mothers
insulin levels | Baseline to 10 months postpartum
  Change in insulin levels in mothers
homeostasis model assessment | Baseline to 10 months postpartum
  Change in homeostasis model assessment calculation in mothers
hemoglobin A1c | Baseline to 10 months postpartum
  Change in hemoglobin A1c in mothers
complete lipid panel | Baseline to 10 months postpartum
  Change in complete lipid panel in mothers
blood pressure | Baseline to 10 months postpartum
  Change in blood pressure in mothers
adiposity | Baseline to 10 months
  Change in adiposity (waist circumference, triceps and subscapular skin folds)in mothers
health behaviors | Baseline to 10 months postpartum
  Change in health behaviors (Health Promoting Lifestyle Profile II, Adult Health Behavior Survey, and Accelerometry for 7 days) in mothers
self-efficacy | Baseline to 10 months postpartum
  Change in self-efficacy in mothers
infant weight status | Birth to 10 months
  weight status (weight-for-length) in children
breastfeeding | Birth to 10 months
  Change in breastfeeding (weeks until stopped breastfeeding, weeks exclusively breastfed, and intensity of breastfeeding) in infants

CONTACTS AND LOCATIONS:
Overall Officials: Diane Berry, PhD, ANP-BC, Principal Investigator — University of North Carolina, Chapel Hill; Alison Stuebe, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC-Rex Health Care, Raleigh, North Carolina
  - WakeMed, Raleigh, North Carolina

REFERENCES:
- [Derived] Stuebe AM, Bonuck K, Adatorwovor R, Schwartz TA, Berry DC. A Cluster Randomized Trial of Tailored Breastfeeding Support for Women with Gestational Diabetes. Breastfeed Med. 2016 Dec;11(10):504-513. doi: 10.1089/bfm.2016.0069. Epub 2016 Oct 26. PMID 27782758
- [Derived] Berry DC, Neal M, Hall EG, Schwartz TA, Verbiest S, Bonuck K, Goodnight W, Brody S, Dorman KF, Menard MK, Stuebe AM. Rationale, design, and methodology for the optimizing outcomes in women with gestational diabetes mellitus and their infants study. BMC Pregnancy Childbirth. 2013 Oct 10;13:184. doi: 10.1186/1471-2393-13-184. PMID 24112417